CLINICAL TRIAL: NCT07298161
Title: Evaluating SleepWhale Drops for Rest & Resilience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 37640
Record Dates: First submitted 2025-12-03; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single arm where participants act as their own control
  Interventions: Dietary Supplement: SleepWhale Natural Sleep Drops

INTERVENTIONS:
Dietary Supplement: SleepWhale Natural Sleep Drops — Broad spectrum hemp extract: 25 mg Broad spectrum hemp extract (CBN): 1.5 mg Proprietary blend of Suntheanine (L-Theanine), GadoMag (Magnesium( Sibelius (Camomile) and M2 (Lion's Mane)

SUMMARY:
30-day study evaluating SleepWhale Natural Sleep Drops (Extra Strength)-formulated to support deeper sleep and better days.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to rigorously evaluate the efficacy of SleepWhale Natural Sleep Drops (Extra Strength), a non-melatonin sleep aid composed of adaptogens and botanicals, in improving sleep quality and daytime well-being. Recognizing the pervasive issues of sleep disturbances including racing thoughts, restless nights, and sluggish mornings, and the growing interest in natural remedies that provide support without the risk of grogginess or dependency, this study aims to provide empirical evidence on the benefits of SleepWhale.

Participants in this trial will incorporate SleepWhale Drops into their nightly routine for a duration of 30 days. Throughout this period, participants are required to complete weekly check-ins utilizing scientifically validated self-report tools. This approach is chosen to emphasize the subjective experience of sleep quality and daytime functioning over metrics that might be collected by sleep trackers or wearable devices, which, while useful, can sometimes lack accuracy and fail to capture the entirety of an individual's sleep experience.

The primary objective of this study is to assess the impact of regular nightly use of SleepWhale Natural Sleep Drops on several key outcomes, including self-reported sleep quality, incidences of sleep disruption, daytime performance, and overall resilience. By focusing on these areas, the study aims to gather meaningful data that reflects the real-world effectiveness of SleepWhale Drops in supporting restful sleep and enhancing daytime productivity and well-being.

Ultimately, by participating in this trial, individuals will not only contribute to their personal health and well-being but also to the larger body of research aimed at validating the effectiveness of SleepWhale Natural Sleep Drops. This study stands as a critical step towards separating trend from truth, offering participants and the wider community real outcomes and insights into the potential of SleepWhale as a natural solution for better sleep and brighter days.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Exclusion Criteria:

* Individuals with Allergies to supplement ingredients
* Individuals on sleep Medication
* Individuals with Gastrointestinal Issues
* Individuals with Skin Conditions
* Individuals Prone to Headaches
* Individuals with Mental Health Conditions
* Pregnant or Breastfeeding Individuals
* Athletes and Competitive Participants
* Individuals with Dependency Issues
* Individuals with Dizziness or Fatigue Issues

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
PROMIS Sleep Disturbance Scale | Change from baseline (Day 1-3) in PROMIS Sleep Disturbance Scale at 4 weeks (Day 28-32)
  The PROMIS Sleep Disturbance Scale is a validated and widely used assessment tool developed as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) initiative. It is designed to measure the severity of sleep disturbances and disruptions experienced by individuals. This scale includes a range of questions that assess the frequency and impact of various sleep-related issues, such as difficulty falling asleep, nighttime awakenings, and restless sleep. Healthcare professionals and researchers rely on this scale to better understand and quantify sleep problems in patients, enabling them to tailor interventions and treatment strategies to address sleep-related concerns effectively.
  Unabbreviated Scale Title Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Scale
  Score Range
  Short Form (e.g., 8a): 8-40
  Score Interpretation
  Higher scores = worse sleep disturbance
  Lower scores indicate better sleep quality
Daytime Sleepiness Perception Scale (DSPS-4) | Change from baseline (Day 1-3) in DSPS-4 at 4 weeks (Day 28-32)
  This survey is designed to measure your perception of daytime sleepiness. Please read each statement carefully and circle the response that best applies to your experience.
  Score Range
  Each item typically scored 0-4 or 1-5
  Total score range (most common): 0-16
  Score Interpretation
  Higher scores = greater perceived daytime sleepiness
  Lower scores indicate better daytime alertness
Fatigue Perception and Impact Survey | Change from baseline (Day 1-3) in FPIS at 4 weeks (Day 28-32)
  The Fatigue Perception and Impact Survey (FPIS) is a specialized questionnaire developed to evaluate the presence, severity, and impact of fatigue on an individual's life. Comprising a series of questions, the survey aims to capture both the subjective experience of fatigue and its consequences across various domains, such as physical, emotional, and social aspects. This tool is commonly used in clinical settings to assess fatigue in patients with various medical conditions, including chronic illnesses and cancer, helping healthcare professionals better understand and address the debilitating effects of fatigue on patients' quality of life. Researchers also employ the FPIS to gather valuable data on fatigue patterns.
  Score Range 0-4 or 1-5 Likert items Total score range 0-50 Score Interpretation Higher score= worse fatigue and greater functional impact Lower score= less perceived fatigue
Resilience Assessment Scale | Change from baseline (Day 1-3) in Resilience Assessment Scale at 4 weeks (Day 28-32)
  This survey aims to evaluate your level of resilience in different situations. Score Range
  0-100 (scaled score)
  Score Interpretation
  Higher scores = greater resilience (better outcome)
  Lower scores indicate reduced psychological resilience

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=37640